CLINICAL TRIAL: NCT00388778
Title: The Effect of Doxycycline 100mg and Doxycycline 20mg in Treatment of Mild and Moderate Acne
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: src-pts-964
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Last update posted 2008-01-23 (Estimated); Status verified 2008-01

CONDITIONS: Acne; Inflammation
MeSH Terms: conditions — Acne Vulgaris; Inflammation | interventions — Doxycycline

INTERVENTIONS:
Drug: Doxycycline

SUMMARY:
The purpose of this study is to compare the safety and efficacy of twice daily subantimicrobial dose doxycycline 20mg with daily doxycycline 100mg in treatment of mild and moderate Acne.

ELIGIBILITY:
Inclusion Criteria:

* Acne

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-10; Study Completion 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: Parviz Toossi, M.D., Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- Skin Research Center, Shaheed Beheshti Medical University, Tehran, Iran